CLINICAL TRIAL: NCT06258941
Title: Supporting High-intensity Interval Training With Mindfulness for Enhancing Childhood Executive Function
Brief Title: Classroom Break, Cognition, and Fitness in Elementary School Children
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Shih-Chun Kao, Assistant Professor, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2024-1588
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers
Keywords: Executive function; Mindfulness; Interval exercise; Children; Fitness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 12-Week Mindful High-Intensity Interval Training (MF-HIIT) (Experimental)
  Interventions: Behavioral: MF-HIIT
- 12-Week High-Intensity Interval Training (HIIT-only) (Active Comparator)
  Interventions: Behavioral: HIIT-only
- 12-Week Mindfulness (MF-only) (Active Comparator)
  Interventions: Behavioral: MF-only
- 12-Week Sedentary Activities (Placebo Comparator)
  Interventions: Behavioral: Sedentary activity

INTERVENTIONS:
Behavioral: MF-HIIT — Two 10-min MF-HIIT sessions every school day during the 12-week intervention period. One session in the morning and one session in the afternoon.
  Arms: 12-Week Mindful High-Intensity Interval Training (MF-HIIT)
Behavioral: HIIT-only — Two 10-min HIIT-only sessions every school day during the 12-week intervention period. One session in the morning and one session in the afternoon.
  Arms: 12-Week High-Intensity Interval Training (HIIT-only)
Behavioral: MF-only — Two 10-min MF-only sessions every school day during the 12-week intervention period. One session in the morning and one session in the afternoon.
  Arms: 12-Week Mindfulness (MF-only)
Behavioral: Sedentary activity — Two 10-min sedentary sessions every school day during the 12-week intervention period. One session in the morning and one session in the afternoon.
  Arms: 12-Week Sedentary Activities

SUMMARY:
The goal of this randomized controlled trial is to learn about the effect of a 12-week school-based intervention combining mindfulness with high-intensity interval training (MF-HIIT), MF-only intervention, and HIIT-only intervention in relative to sedentary activities on executive function (EF) in 8-12 years old children. The main question it aims to answer is whether a 12-week school-based MF-HIIT intervention has larger beneficial effect on EF performance than that following a 12-week school-based MF-only and HIIT-only in relative to the sedentary activities.

Multiple cohorts of participants will be recruited to participate this one-semester study, including the pretest, intervention, and posttest phases.

During the pretest phase, participants an their parents will complete the following

1. Kaufman Brief Intelligence Test (KBIT) to assess intelligence quotient
2. Fitnessgram test to assess aerobic capacity, muscle endurance, flexibility, and body mass index
3. Child and Adolescent Mindfulness Measure (CAMM) questionnaire to assess dispositional mindfulness
4. Computerized tasks to assess EF
5. Parent-reported demographic and health information

Following the pretest phase, participants will receive the 12-week classroom-based intervention, with the classroom as the intervention unit.

Following the intervention and during the posttest phase, participants will complete the fitness, measures, EF measures, and dispositional mindfulness measure again.

Researcher will compare the EFn outcome measures following the MF-HIIT, MF-only, and HIIT-only interventions with the sedentary activity intervention to see if MF and HIIT has beneficial effects on children's EF.

Further, researcher will compare the EF measures following the MF-HIIT compared with MF-only and HIIT-only interventions to see if combining MF with HIIT has greater beneficial effects on children's EF than MF and HIIT alone.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8-12 years old
* Intelligence Quotient ≥ 70
* Capable of performing exercise based on pre-participation health screening
* No formal diagnosis of neurological diseases (e.g., epilepsy)

Exclusion Criteria:

* Age outside of the range of 8-12 years old
* Intelligence Quotient < 70
* No capable of performing exercise based on pre-participation health screening
* Has formal diagnosis of neurological diseases (e.g., epilepsy)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 352 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Inhibition speed | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Inhibition speed will be assessed by the response time (ms) during a child-friendly flanker task.
Inhibition accuracy | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Inhibition accuracy will be assessed by the response accuracy (percent) during a child-friendly flanker task.
Updating speed | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Updating speed will be assessed by the response time (ms) during a child-friendly n-back task.
Updating accuracy | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Updating accuracy will be assessed by the response accuracy (percent) during a child-friendly n-back task.
Shifting speed | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Shifting speed will be assessed by the response time (ms) during a child-friendly switching task.
Shifting accuracy | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Shifting accuracy will be assessed by the response accuracy (percent) during a child-friendly switching task.

SECONDARY OUTCOMES:
Aerobic capacity | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Aerobic capacity will be assessed by the Progressive Aerobic Cardiovascular Endurance Run (PACER) test
Upper body muscle endurance | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Upper body muscle endurance will be assessed by the push-ups test
Core body muscle endurance | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Core body muscle endurance will be assessed by the curl-ups test
Flexibility | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Flexibility will be assessed by the back-saver sit and reach test
Body composition | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  body composition will be assessed by the body mass index computed as weight (kg) / (height [m] * height [m])
Dispositional mindfulness | At the baseline (1-2 weeks) before intervention starts and after (1-2 weeks) the intervention ends
  Dispositional mindfulness will be assessed by the Child and Adolescent Mindfulness Measure questionnaire (CAMM). The questionnaire has 10 items and requires the respondents to rating each item using a 5-point likert scale from 0 (Never True) to 4 (Always True). Higher summed scores indicate higher levels of mindfulness

CONTACTS AND LOCATIONS:
Locations (1):
- Pioneer Elementary School, Royal Center, Indiana, United States